CLINICAL TRIAL: NCT00470678
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Ranibizumab (0.5 mg) in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration Over 12 Months
Brief Title: EXTEND III - Efficacy and Safety of Ranibizumab in Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002A2304
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Choroidal Neovascularization; Age-Related Macular Degeneration
Keywords: Age-related; macular; degeneration; AMD; Ranibizumab; Anti-VEGF; choroidal; neovascularization; CNV; Asian patients; Korea; Taiwan; associated
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration; Neovascularization, Pathologic | interventions — Ranibizumab

ARMS (1):
- 1 (Experimental): Ranibizumab
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab
  Other Names: Lucentis, RFB002

SUMMARY:
This study will evaluate efficacy and safety for monthly ranibizumab 0.5 mg intravitreal injections in Asian patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Asian patients 50 years of age or greater.
* Patients with primary or recurrent subfoveal CNV secondary to AMD, including those with predominantly classic, minimally classic or active occult lesions with no classic component.
* Patients who have a BCVA score between 73 and 24 letters (approximately 20/40 to 20/320 Snellen equivalent), inclusively, in the study eye.
* Total area of CNV (including both classic and occult components) encompassed within the lesion must be >= 50% of the total lesion area
* Total lesion area must be <= 12 disc areas

Exclusion Criteria:

* Patients who have in the fellow eye a Snellen equivalent below 20/200
* Presence of angioid streaks, presumed ocular histoplasmosis syndrome, myopia (exceeding -8 diopters), or CNV secondary to causes other than AMD in the study eye
* Subfoveal fibrosis or atrophy in the study eye
* Total area of CNV (including both classic and occult components) encompassed within the lesion must be >= 50% of the total lesion area
* Total lesion area must be <= 12 disc areas
* Vitreous hemorrhage, retinal tear or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye.
* Active, or history of, ocular inflammation or infection in the study eye within the last 30 days prior to screening.
* Uncontrolled glaucoma in the study eye
* Treatment in the study eye with verteporfin, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, submacular surgery, or transpupillary thermotherapy within 30 days prior to screening
* Previous treatment with anti-angiogenic drugs (pegaptanib, ranibizumab, bevacizumab, anecortave acetate, corticosteroids, protein kinase C inhibitors, squalamine, siRNA, VEGF-Trap etc.) for neovascular AMD in the study eye. Treatment of the fellow eye is permitted if administered > 30 days before screening.
* History of intraocular surgery in the study eye including pars plana vitrectomy, except for uncomplicated cataract surgery more than 60 days prior to screening
* History of YAG laser posterior capsulotomy in the study eye within 30 days prior to screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) from Baseline, Month 4 and Month 12 as assessed with ETDRS (Early Treatment for Diabetic Retinopathy Study)-like charts at a distance of four meters | Baseline, Month 4 and Month 12

SECONDARY OUTCOMES:
Changes in the retinal structure from baseline as assessed by fundus photography and fluorescein angiography, Month 4 and Month 12 | Month 4 and Month 12
Safety by rates of adverse events and serious adverse events, ophthalmic examinations, tonometry, and vital signs, baseline, Month 4, Month 6 and Month 12 | Baseline, Month 4, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis
Locations (6):
- South Korea (3):
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Pusan
  - Novartis Investigative site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative site, Taipei

REFERENCES:
- [Result] Kwon OW, Lee FL, Chung H, Lai CC, Sheu SJ, Yoon YH; EXTEND III study group. EXTEND III: efficacy and safety of ranibizumab in South Korean and Taiwanese patients with subfoveal CNV secondary to AMD. Graefes Arch Clin Exp Ophthalmol. 2012 Oct;250(10):1467-76. doi: 10.1007/s00417-012-1970-3. Epub 2012 Mar 2. PMID 22382503